CLINICAL TRIAL: NCT04295096
Title: Collection of Peripheral Blood Mononuclear Cells From Healthy Subjects for the Development of Cellular Immunotherapy Product
Brief Title: Collection of PBMCs From Healthy Subjects for the Development of Cellular Immunotherapy Product
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Zhu (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhu, Chief Physician, Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai
Organization: Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BM2L201909
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Healthy Subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Other): Healthy donor
  Interventions: Device: Peripheral blood mononuclear cell apheresis

INTERVENTIONS:
Device: Peripheral blood mononuclear cell apheresis — Peripheral blood mono-nuclear cell donation for tumor immunotherapy study of Universal CAR-T cells

SUMMARY:
Title: Collection of Peripheral Blood Mononuclear Cells (PBMCs) From Healthy Subjects for the Development of Cellular Immunotherapy Product

Background:

CAR-T therapies are being developed that utilize modified immune cells to fight tumors. 'Off-the-shelf' allogeneic CAR-T technology has better efficacy and more promising clinical applications. Investigators want to use the cells of healthy subjects to perform the studies. To accomplish this, they are collecting PBMCs through apheresis.

Objectives:

To collect PBMCs from healthy subjects for product development for cell Immunotherapies.

DETAILED DESCRIPTION:
Background:

Autologous chimeric antigen receptor (CAR) T cells have changed the therapeutic landscape in haematological malignancies. Nevertheless, the use of allogeneic CAR T cells from donors has many potential advantages over autologous approaches, such as the immediate availability of cryopreserved batches for patient treatment, possible standardization of the CAR-T cell product, time for multiple cell modifications, redosing or combination of CAR T cells directed against different targets, and decreased cost using an industrialized process. The T cells currently used for CAR-T cell manufacturing are mainly derived from peripheral blood mono-nuclear cells (PBMCs) .The manufacture of allogeneic CAR T cells from PBMCs collected from healthy donors is associated with the ability to make multiple vials from a single apheresis product. Allogeneic CAR T cells are created from healthy donors, they are generated from immune cells that have not been impacted by the immune effects of cancer or by exposure to chemotherapeutic agents, in contrast to autologous T cells from patients. The selection of donors on the basis of their immune characteristics is likely to be a key factor in decreasing the heterogeneity of the final cell product

Objectives:

* To produce allogeneic CAR T cells with different targets and other cell products by using PBMCs from healthy subjects.
* To develop and optimize the methodology for the response or quality determination of cell Immunotherapy products.

Design:

All subjects are required to sign a written informed consent form for the study. After the signing of informed consent form, participants will be screened with a series of vital signs, physical examinations and laboratory tests. Demographic data and medical history of the subjects will also be documented. In addition, 30 mL peripheral venous blood sample will be collected to evaluate the biological characteristics of each subject. Participants will undergo a routine blood test within 24 hours before the apheresis to reconfirm their eligibility and 3-5 mL blood samples are to be drawn for the development of detection methods of cell-based immunotherapy. Subjects who meet all the inclusion criteria and do not meet any exclusion criteria are qualified to donate peripheral blood mono-nuclear cells (PBMCs) by means of apheresis. 6×10[9] of cells for each healthy person are preferred. 172 healthy subjects are to be enrolled through the whole study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age
* Male≥50 kg, female≥45 kg with 18.5≤ BMI ≤30
* Subject has provided informed consent

Exclusion Criteria:

* Subject has respiratory diseases, circulatory system diseases, digestive system diseases, urinary system diseases, hematological system diseases, autoimmune diseases, endocrine disorders or metabolic disorders;
* Subject has nervous system diseases, mental illness, Creutzfeldt-Jakob disease or those with a family history, or those treated with tissue or tissue derivatives that may be derived from Creutzfeldt-Jakob infected people;
* Subject has chronic skin diseases, especially infectious, allergic or inflammatory systemic skin diseases;
* Subject has allergic diseases or recurrent allergies;
* Malignant tumors or health-affecting benign tumors;
* Twice or more times of blood pressure measurement exhibit (except for white coat hypertension): systolic blood pressure < 90 or ≥ 140 Millimeter of mercury (mm Hg), or diastolic blood pressure < 60 or ≥ 90 mm Hg, or pulse pressure < 30 mm Hg, heart rate: < 60 beats/min or >100 beats/min;
* Laboratory tests: hemoglobin: male <120 g/L, female <115 g/L, or liver and kidney laboratory result >1.5x upper limit of normal with clinical significant, or abnormal12-lead ECG with clinical significant, or abnormal abdominal B-mode ultrasound with clinical significant, or abnormal chest X-ray with clinical significant, and T cell detection of tuberculosis infection is over the limit or positive;
* Abnormal lymphocyte subset panel test result with clinical significance (Lymphs%, CD3+, CD3+CD4+, CD3+CD8+, CD3-CD16+CD56+,CD19+) ;
* Hepatitis B surface antigen positive, hepatitis B virus (HBV) DNA positive, hepatitis B e antigen positive, hepatitis C antibody positive, Treponema pallidum antibody positive ,human immunodeficiency virus antibody positive, human T-cell lymphotrophic virus antibody positive, Epstein-Barr virus positive, or COVID-19 nucleic acid positive ;
* Recipient of organ transplant;
* Received any major organ resection such as stomach, kidney, spleen and lung;
* Subject has transfusion-associated infectious diseases;
* Minor surgery within 3 months, such as appendectomy and recovered ophthalmic surgery; Major surgery within l 1 year, such as surgical treatment for gynecological benign tumors or superficial benign tumors;
* Pregnant, or have an abortion within l 6 months, childbirth within 1 year;
* Upper respiratory infection recovered within 1 week, or pneumonia recovered within 3 months;
* Acute pyelonephritis-recovered within 3 months, or urinary calculi onset;
* Injured or wound-contaminated by equipment contaminated by blood or tissue fluids, or has a tattoo within 1 year;
* Received whole blood and blood component transfusion within 1 year;
* Received the last vaccination of live attenuated vaccines such as measles, mumps, or polio within 2 weeks, or the last vaccination of rubella live vaccine, human rabies vaccine, live attenuated Japanese encephalitis vaccine within 4 weeks;
* Received the last vaccination of rabies vaccines after being bitten by an animal within 1 year;
* Received the last vaccination of antitoxin or immune serum injection within 4 weeks, or those who received the last vaccination of hepatitis B human immunoglobulin injection within 1 year;
* Participated in a clinical trials within 1 month; it should be discussed case by base if investigational product used.
* Those who are considered by the investigator as unsuitable for participating in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Collect blood samples | 2 years
  Collect blood samples (whole blood and PBMC) from healthy subjects for the Development of Cellular Immunotherapy Product.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, M.D., Principal Investigator — Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai
Locations (1):
- Zhaxin Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No